CLINICAL TRIAL: NCT00224393
Title: Phase II Trial of Enbrel in Patients With Primary Systemic Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC018A
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Primary Systemic Amyloidosis
Keywords: Amyloidosis; Enbrel
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis; Amyloidosis | interventions — Etanercept

INTERVENTIONS:
Drug: Enbrel

SUMMARY:
The purpose of this study is to evaluate the efficacy of Enbrel in patients with primary systemic Amyloidosis.

DETAILED DESCRIPTION:
The primary goal of this study is to evaluate the efficacy of Enbrel in patients with primary systemic amyloidosis using a one-stage, phase II study design with an interim analysis. This study will also assess survival and progression times, symptom relief, and toxicity associated with Enbrel in primary systemic amyloidosis patients. Two groups of patients with very different risk profiles can be identified with respect to this disease. Patients with symptomatic cardiac disease and/or at least two involved organs ar at high risk and historically have a median survival less than six months. Patients without these conditions have a significantly better prognosis. Both subgroups will be studied in the present study, and essentially two phase-II clinical trials, one for each subgroup, will be run in parallel.

ELIGIBILITY:
Inclusion Criteria:

* >=18 years of age.
* Laboratory values obtained <=14 days prior to registration.
* No limitation on the cardiac ejection fraction
* Bilirubin <3 mg/dL
* Absolute neutrophil count >=500/microliters
* Histochemical diagnosis of amyloidosis as based on detection by polarizing microscopy of green bi-refringent material in Congo red-stained tissue specimens or characteristic electron microscopy appearance.
* Demonstrable M-protein in the serum/urine or clonal population of plasma cells in the bone marrow or immunohistochemical stain with anti-light chain anti-sera of amyloid fibrils.
* ECOG performance status 0, 1, 2, or 3.
* Symptomatic organ involvement with amyloid to justify therapy. This could include liver involvement, cardiac involvement, renal involvement, peripheral neuropathy, or soft tissue involvement. Must have more than purpura or carpal tunnel syndrome.
* Previously treated or untreated. No limit to prior therapy provided there is adequate residual organ function.
* Ability to provide informed consent.
* Ability to self-inject medication or have a caregiver who can administer the drug.

Exclusion Criteria:

* Amyloid-specific syndrome, such as, carpal tunnel syndrome or skin purpura as only evidence of disease. The finding of vascular amyloid only in a bone marrow biopsy specimen or in a plasmacytoma is not indicative of systemic amyloidosis.
* Presence of non-AL amyloidosis.
* Melphalan or other alkylating agents, high-dose dexamethasone or alpha interferon <=4 weeks prior to registration.
* Concurrent use of corticosteroids, but patients may be on chronic steroids if they are being given for disorders other than amyloid, i.e., adrenal insufficiency, rheumatoid arthritis, etc.
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, abstinence, etc.)
* Uncontrolled infection.
* Clinically overt multiple myeloma (monoclonal BMPC >30%), and at least one of the following:

  * Bone lesions
  * Hypercalcemia
* Active malignancy with the exception of adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2001-02; Study Completion 2005-08-31 (Actual)

PRIMARY OUTCOMES:
clinical efficacy

SECONDARY OUTCOMES:
Duration of response and time to progression
Evaluate overall survival
Identify prognostic factors
Evaluate qualitative and quantitative toxicities of Enbrel

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad A Hussein, MD, Principal Investigator — The Cleveland Clinic; John A Lust, MD, PhD, Study Chair — Mayo Clinic